CLINICAL TRIAL: NCT04527913
Title: Interdental Plaque Reduction After Use of Different Devices in Patients With Periodontitis: a Randomized Clinical Trial
Brief Title: Interdental Plaque Reduction and Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Full Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Periobrush
Record Dates: First submitted 2020-08-12; First posted 2020-08-27 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Single-centre randomized, parallel design, clinical trial with a five-week follow-up
Who Masked: Investigator, Outcomes Assessor
Masking Description: Center will enroll probands, assigning a unique study subject number and allocating an opaque randomization envelope.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Experimental): 15 patients receiving oral hygiene instructions as determined by their group allocation (use of manual toothbrush alone)
  Interventions: Procedure: One session of professional supragingival scaling and polishing; Procedure: Oral Hygiene Instruction (OHI)
- Test group 1 (Experimental): 15 patients receiving oral hygiene instructions as determined by their group allocation (manual toothbrush plus dental floss)
  Interventions: Behavioral: Interdental Oral Hygiene Instruction (Int-OHI); Procedure: One session of professional supragingival scaling and polishing; Procedure: Oral Hygiene Instruction (OHI)
- Test group 2 (Experimental): 15 patients receiving oral hygiene instructions as determined by their group allocation (manual toothbrush plus interdental brushes)
  Interventions: Behavioral: Interdental Oral Hygiene Instruction (Int-OHI); Procedure: One session of professional supragingival scaling and polishing; Procedure: Oral Hygiene Instruction (OHI)
- Test group 3 (Experimental): 15 patients receiving oral hygiene instructions as determined by their group allocation (manual toothbrush plus rubber interdental picks)
  Interventions: Behavioral: Interdental Oral Hygiene Instruction (Int-OHI); Procedure: One session of professional supragingival scaling and polishing; Procedure: Oral Hygiene Instruction (OHI)

INTERVENTIONS:
Behavioral: Interdental Oral Hygiene Instruction (Int-OHI) — Int-OHI will be given focusing on the interdental device of the allocated group for each patient and will be given only once at timepoint T-7. No further formal Int-OH instructions will be given, unless specifically asked by the patient.
  Int-OHI will be delivered by trained dental hygienist/periodontist.
  Arms: Test group 1; Test group 2; Test group 3
Procedure: One session of professional supragingival scaling and polishing — A session of professional supragingival scaling and polishing: instrumentation will be performed by a trained dental hygienist/periodontist with great care in performing exclusively coronal maneuver. No instrumentation or exploring of the gingival crevice/ sulcus will be performed.
Procedure: Oral Hygiene Instruction (OHI) — OHI will be given focusing on manual toothbrushing and will be given only once at timepoint T-7. No further formal OH instructions will be given, unless specifically asked by the patient.
  OHI will be delivered by trained dental hygienist/periodontist.

SUMMARY:
To determine the efficacy of four different oral hygiene protocols involving adjunctive interdental cleaning devices in periodontal patients in terms of plaque and gingival inflammatory scores.

DETAILED DESCRIPTION:
Patients included in the study will undergo a thorough clinical examination aiming at collecting all the data desired: periodontal parameters of Probing Pocket Depth (PPD), presence of recession of the gingival margin (Rec) and full mouth plaque score (FMPS) will be recorded on six sites/tooth by a single calibrated examiner using a University of North Carolina (UNC) 15-mm periodontal probe by a calibrated examiner blind to group allocation.

Gingival index (GI) and angulated bleeding score (AngBS) will be recorded at four sites/tooth.

For GI the following scale will be used:

0 normal appearance of gingiva, no bleeding, no inflammation;

1. slight change and moderate edema with slight change in texture, no bleeding, mild inflammation;
2. redness hypertrophy, or edema and glazing, bleeding on probing, moderate inflammation;
3. marked redness, hypertrophy, or edema, ulceration, spontaneous bleeding, severe inflammation.

For AngBS the following scale will be used:

0: no bleeding;

1. bleeding upon probe stimulation;
2. spontaneous bleeding

Consequently, interdental plaque score (IPS), interdental gingival index (IGI), and interdental angulated bleeding score (IAngBI) will be calculated.

Patients will be followed through a five-week period. The timepoints will be the following: T -7 (oral hygiene instructions), T0 (professional supragingival scaling and polishing), T14, T28.

ELIGIBILITY:
Inclusion Criteria:

* males or females of age range between 18 and 70 years,
* good health status,
* presence of at least 20 natural teeth
* residual periodontal pockets with PPD≥4mm, in need of specific oral hygiene regimen.

Exclusion Criteria:

* pregnancy or breast-feeding,
* indication to antibiotic therapy prior to treatment,
* chronic infections,
* systemic diseases (including cardiovascular, pulmonary, cerebral, and metabolic diseases),
* not willing to give a consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
FMPS Full-mouth plaque score (FMPS) | Measured at: Baseline, at 1 week, at 3 weeks, and at 5 weeks
  Changes in FMPS, measured orally through clinical examination. Unit of measure: N

SECONDARY OUTCOMES:
Pocket probing depth (PPD) | Measured at Baseline and at 5 weeks
  Changes in PPD, measured orally through clinical examination. Unit of measure: mm
Recession of the gingival margin (REC) | Measured at Baseline and at 5 weeks
  Changes in REC, measured orally through clinical examination. Unit of measure: mm
Clinical attachment level (CAL) | Measured at Baseline and at 5 weeks
  Changes in CAL, measured orally through clinical examination. Unit of measure: mm
Gingival Index (GI) | Measured at: Baseline, at 1 week, at 3 weeks, and at 5 weeks
  Changes in GI, measured orally through clinical examination. Unit of measure: scale from 0 (normal) to 3 (Marked redness, hypertrophy, or edema, ulceration)
Angulated bleeding score (AngBS) | Measured at: Baseline, at 1 week, at 3 weeks, and at 5 weeks
  Changes in AngBS, measured orally through clinical examination. Unit of measure: scale from 0 (no bleeding), 1 (bleeding upon probe stimulation) to 2 (spontaneous bleeding).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided